CLINICAL TRIAL: NCT00544037
Title: Extension Study of the BENEFIT (304747) and BENEFIT Follow-up (305207) Studies to Further Evaluate the Progress of Patients With First Demyelinating Event Suggestive of Multiple Sclerosis
Brief Title: BENEFIT Extension Study
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Global Medical Affairs Therapeutic Area Head, Byer Healthcare AG
Other Study IDs: 91713; 311129 (Other: Company internal)
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Population of Benefit Studies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Standard Therapy for Multiple Sclerosis

SUMMARY:
To assess the long-term effects of early therapeutic intervention, i.e. within two years following a first clinical demyelinating event suggestive of MS.

ELIGIBILITY:
Inclusion Criteria:

* All patients randomized and treated at least once in study 304747

Exclusion Criteria:

* Medical, psychiatric or other conditions that compromise the patient's ability to understand the purpose of the study

Ages: 23 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This observational study may include all patients who were randomized into and treated at least once in the BENEFIT study 304747, inclusive of patients who prematurely discontinued study participation in either study 304747 or study 305207, and patients who did not transfer from study 304747 to study 305207.
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2007-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To obtain further clinical data of patients with a first demyelinating event suggestive of Multiple Sclerosis enrolled in the BENEFIT Study | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (18):
- Many Locations, Austria
- Many Locations, Belgium
- Many Locations, Canada
- Many Locations, Czechia
- Many Locations, Denmark
- Many Locations, Finland
- Many Locations, France
- Many Locations, Germany
- Many Locations, Hungary
- Many Locations, Israel
- Many Locations, Italy
- Many Locations, Netherlands
- Many Locations, Norway
- Many Locations, Poland
- Many Locations, Slovenia
- Many Locations, Spain
- Many Locations, Sweden
- Many Locations, Switzerland

REFERENCES:
- [Derived] Nagtegaal GJ, Pohl C, Wattjes MP, Hulst HE, Freedman MS, Hartung HP, Miller D, Montalban X, Kappos L, Edan G, Pleimes D, Beckman K, Stemper B, Polman CH, Sandbrink R, Barkhof F. Interferon beta-1b reduces black holes in a randomised trial of clinically isolated syndrome. Mult Scler. 2014 Feb;20(2):234-42. doi: 10.1177/1352458513494491. Epub 2013 Jul 10. PMID 23842212